CLINICAL TRIAL: NCT01995240
Title: Functional Magnetic Resonance Imaging of Pancreatic Cancer: a Feasibility and Reproducibility Study
Acronym: REMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, H.W.M. van Laarhoven, M.D., Ph.D., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NL40501.018.12
Record Dates: First submitted 2013-11-21; First posted 2013-11-26 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2017-03

CONDITIONS: Pancreatic Cancer
Keywords: pancreatic cancer; MRI; reproducibility; optimalization
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — gadobutrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Optimization (Experimental): For optimization of the protocol patients will undergo one DCE-MRI (Gadobutrol), T2* MRI and DWI MRI scan.
  Interventions: Drug: Gadobutrol
- Reproducibility (Experimental): For determination of the reproducibility patients will undergo two DCE-MRI (Gadobutrol), T2* MRI and DWI MRI scans within one week.
  Interventions: Drug: Gadobutrol

INTERVENTIONS:
Drug: Gadobutrol — 0.1 ml/kg Gadovist is administered at 5 ml/s followed by a 15 ml saline flush
  Other Names: Gadovist

SUMMARY:
Novel predictive markers are needed to determine treatment efficacy in pancreatic cancer at an early stage. Preferably, these markers could be determined non-invasively and provide insight into the biology of pancreatic cancer. Several MR techniques can serve for this purpose. However, optimalisation of these techniques is needed and their reproducibility should be assessed.

DETAILED DESCRIPTION:
Background of the study:

Novel predictive markers are needed to determine treatment efficacy in pancreatic cancer at an early stage. Preferably, these markers could be determined non-invasively and provide insight into the biology of pancreatic cancer. Several MR techniques can serve for this purpose. However, optimalisation of these techniques is needed and their reproducibility should be assessed.

Objective of the study:

To optimize DCE-MRI, T2* MRI and DWI in pancreatic cancer at 3T and investigate its reproducibility.

Study design:

In the first part of the study, patients with pancreatic cancer will undergo an MR measurement protocol once at 3T, to optimize MR techniques (DCE-MRI, T2* MRI and DWI). In the second part of the study, to assess reproducibility patients will undergo the MR measurement protocol twice within one week before start of any treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pancreatic tumors, with histological or cytological proof of adenocarcinoma or a high suspicion on CT imaging.
* Any tumor with a size ≥ 1cm
* WHO-performance score 0-2
* Written informed consent

Exclusion Criteria:

* Any psychological, familial, sociological or geographical condition potentially hampering adequate informed consent or compliance with the study protocol.
* Contra-indications for MR scanning, including patients with a pacemaker, cochlear implant or neurostimulator; patients with non-MR compatible metallic implants in their eye, spine, thorax or abdomen; or an aneurysm clip in their brain; patients with severe claustrophobia.
* Renal failure (GFR < 30 ml/min) hampering safe administration of Gadolinium containing MR contrast agent.
* For the reproducibility part of the protocol: surgery, radiation and/or chemotherapy foreseen within the timeframe needed for MRI scanning.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Reproducibility of DCE, T2* and DWI MRI in pancreatic cancer. | Within 1 week
  To assess reproducibility, 15 patients will undergo the MR measurement protocol twice within one week before start of any treatment.
  Reproducibility of; DWI: mean ADC of the whole tumor. DCE: mean Ktrans of the whole tumor. T2*: average value of the whole tumor.

SECONDARY OUTCOMES:
Compare in vivo measurements of tumor vascularity, hypoxia and stroma using DCE-MRI, T2* MRI and DWI with immunohistochemically determined markers of vascularity, hypoxia and stroma in pancreatic tumor tissue | Within 1 week
  In those patients for whom tumor tissue is available which has not been treated with radiation or chemotherapy, DCE-MRI, T2* MRI and DWI will be compared with immunohistochemical markers of vascularity, hypoxia and stroma (e.g. CD-31, HIF1-alfa, CA9, GLUT1, PAI-1, VEGF, anti-SMA).
To explore the relation between in vivo measurements of tumor vascularity, hypoxia and stroma using DCE-MRI, T2* MRI and DWI and treatment outcome. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: H WM van Laarhoven, M.D., Ph.D., Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academic Medical Center, Amsterdam, Netherlands